CLINICAL TRIAL: NCT01346267
Title: Randomized Controlled Trial of Acupressure to Control Chemotherapy-Induced Nausea (CIN) in Children Receiving Highly Emetogenic Chemotherapy
Brief Title: Acupressure in Controlling Nausea in Young Patients Receiving Highly Emetogenic Chemotherapy
Acronym: SCUSF1202
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SCUSF 1202; SCUSF-1202 (Other: SunCoast CCOP Research Base); Previously COG-ACCL1032 (Other: Children's Oncology Group); 5U10CA081920 (NIH)
Record Dates: First submitted 2011-04-29; First posted 2011-05-02 (Estimated); Results first posted 2021-06-25 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2017-10

CONDITIONS: Central Nervous System Tumor, Pediatric; Chemotherapy-induced Nausea and Vomiting; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; unspecified childhood solid tumor; childhood central nervous system embryonal tumor; childhood central nervous system germ cell tumor; childhood central nervous system germinoma; childhood central nervous system mixed germ cell tumor; childhood central nervous system teratoma; childhood central nervous system yolk sac tumor; childhood mixed glioma; childhood oligodendroglioma; untreated childhood brain stem glioma; untreated childhood visual pathway and hypothalamic glioma; untreated childhood visual pathway glioma; childhood high-grade cerebellar astrocytoma; childhood high-grade cerebral astrocytoma; childhood low-grade cerebellar astrocytoma; childhood low-grade cerebral astrocytoma; untreated childhood cerebellar astrocytoma; untreated childhood cerebral astrocytoma; untreated childhood subependymal giant cell astrocytoma; childhood ependymoblastoma; untreated childhood medulloblastoma; untreated childhood pineoblastoma; childhood choroid plexus tumor; childhood craniopharyngioma; childhood supratentorial ependymoma; childhood supratentorial primitive neuroectodermal tumor; childhood medulloepithelioma; childhood infratentorial ependymoma; newly diagnosed childhood ependymoma; childhood meningioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Vomiting; Nausea; Oligodendroglioma; Astrocytoma; Choroid Plexus Neoplasms; Meningioma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I- Real Acupressure bands (Experimental): Patients wear Sea-Band acupressure wristbands on each wrist beginning approximately 30 minutes prior to the first cisplatin-containing chemotherapy course and continually for 24 hours after the last chemotherapy dose (acute phase), and for a maximum of 7 days or until the next chemotherapy course starts (delayed phase). Patients are allowed to take bands off intermittently (up to 4 times a day, for no more than 15 minutes each time) to relieve pressure or to bathe. Patients also receive standard of care anti-emetic prophylaxis comprising granisetron, ondansetron, or dexamethasone during chemotherapy according to institutional or physician preference.
  Interventions: Procedure: Real Acupressure Band
- Arm II- Placebo Acupressure Bands (Sham Comparator): Patients wear placebo wristbands on each wrist and receive standard of care anti-emetic prophylaxis during chemotherapy as patients in arm I.
  Interventions: Procedure: Placebo Acupressure Band

INTERVENTIONS:
Procedure: Real Acupressure Band — Acupressure wristband
  Arms: Arm I- Real Acupressure bands
Procedure: Placebo Acupressure Band — Sham wristband
  Other Names: sham intervention
  Arms: Arm II- Placebo Acupressure Bands

SUMMARY:
RATIONALE: Acupressure wristbands may prevent or reduce nausea and caused by chemotherapy. It is not yet known whether standard care is more effective with or without acupressure wristbands in controlling acute and delayed nausea.

PURPOSE: This randomized phase III trial is studying how well acupressure wristbands work with or without standard care in controlling nausea in young patients receiving highly emetogenic chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the control of chemotherapy-induced nausea (CIN) in the acute phase provided by a 5-HT3 antagonist combined with acupressure versus placebo acupressure in children 4 to 18 years of age being treated with chemotherapy including cisplatin ≥ 50 mg/m2/dose, ifosfamide plus etoposide/doxorubicin, or cyclophosphamide plus an anthracycline.

Secondary

* To compare the control of CIN in the delayed phase provided by a 5-HT3 antagonist combined with acupressure versus placebo acupressure in children 4 to 18 years of age being treated with chemotherapy including cisplatin ≥ 50 mg/m2/dose, ifosfamide plus etoposide/doxorubicin, or cyclophosphamide plus an anthracycline.
* To compare the control of chemotherapy-induced vomiting and retching (CIV) in the acute and delayed phases provided by a 5-HT3 antagonist combined with acupressure versus placebo acupressure in children 4 to 18 years of age being treated with chemotherapy including cisplatin ≥ 50 mg/m2/dose, ifosfamide plus etoposide/doxorubicin, or cyclophosphamide plus an anthracycline.

OUTLINE: This is a multicenter study. Patients are stratified according chemotherapy regimen and anti-emetic Regimen 5-HT3 agonists (ondansetron or granisetron.) Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients wear Sea-Band acupressure wristbands on each wrist beginning approximately 30 minutes prior to the first cisplatin-containing chemotherapy course and continually for 24 hours after the last chemotherapy dose (acute phase), and for a maximum of 7 days or until the next chemotherapy course starts (delayed phase). Patients are allowed to take bands off intermittently (up to 4 times a day, for no more than 15 minutes each time) to relieve pressure or to bathe. Patients also receive standard of care anti-emetic prophylaxis comprising granisetron, ondansetron, or dexamethasone during chemotherapy according to institutional or physician preference.
* Arm II: Patients wear placebo wristbands on each wrist and receive standard of care anti-emetic prophylaxis during chemotherapy as patients in arm I.

Patients, parents, or guardians are instructed to complete an impatient and an outpatient diaries on nausea severity and the time of each emetic episode. Patients, parents, or guardians also complete a questionnaire about acupressure at the end of the study.

ELIGIBILITY:
INCLUSION CRITERIA:

* 4 to 18 years of age, inclusive. The patient's cognitive ability must be considered by a parent or healthcare professional to be at least at a 4 year-old level.
* Newly diagnosed (i.e., not relapsed) with any malignancy.
* Patients are not required to be registered on a COG therapeutic trial.
* The patient's current chemotherapy treatment plan must include at least 1 course of

  * cisplatin at ≥ 50 mg/m2/dose or
  * ifosfamide plus etoposide or doxorubicin or
  * cyclophosphamide plus an anthracycline.
* Patients may have previously received other chemotherapy.
* The patient's current treatment plan must include an anti-emetic regimen with either ondansetron or granisetron on a scheduled basis. Patients may also receive dexamethasone for antiemetic prophylaxis during the acute phase at the discretion of the treating physician. Patients ≥ 12 years old may also receive aprepitant in conjunction with dexamethasone for antiemetic prophylaxis at the discretion of the treating physician.
* Patients needing anti-emetic treatment for breakthrough nausea/vomiting may also receive anti-emetic agents on an as needed (PRN) basis.
* The patient (parent/guardian) must be English-speaking (i.e., able to read and speak in English) since the PeNAT has been validated only in English.
* All patients and/or their parents or legal guardians must sign a written informed consent (patient assent is also recommended when applicable according to each institution's policy).

EXCLUSION CRITERIA:

* Prior history of acupressure use.
* Scheduled use of antiemetic agents other than ondansetron, granisetron, dexamethasone or aprepitant. Patients may receive other antiemetic agents PRN for breakthrough nausea/vomiting but not on a scheduled basis

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 187 (Actual)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Williams McLean, MD, Study Chair — Wake Forest University Health Sciences; Lee Dupuis, PhD, Study Chair — The Hospital for Sick Children
Locations (25):
- United States (24):
  - Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - A I duPont Hospital for Children, Wilmington, Delaware
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital of Southwest Florida at Lee Memorial, Fort Myers, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Palms West Hospital, Loxahatchee Groves, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Kapiolani Medical for Women and Children, Honolulu, Hawaii
  - Ochsner Clinic Foundation New Orleans, New Orleans, Louisiana
  - Dana Farber Cancer Institute at Boston Children's Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Mercy Children's Hospital, Toledo, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - CHRISTUS Santa Rosa Children's Hospital, San Antonio, Texas
  - Methodist Healthcare System of San Antonio, San Antonio, Texas
  - Scott & White Pediatrics, Temple, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands
Started | 93 | 94
Completed | 70 | 67
Not Completed | 23 | 27

BASELINE CHARACTERISTICS:
Population: 93 participants were allocated to acupressure bands and 83 received the intervention. 94 participants were allocated to the placebo bands and 82 received the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.5 (4.3) | 12.9 (4.2) | 12.7 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 46 | 50 | 96
Diagnosis [Count of Participants; unit: Participants]
  Osteosarcoma | 16 | 17 | 33
  Hodgkin Lymphoma | 20 | 29 | 49
  Ewing Sarcoma | 9 | 6 | 15
  Other | 38 | 30 | 68

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Treatment on CIN During Acute Phase of Chemotherapy
Description: CIN = Chemotherapy-Induced Nausea. The acute phase began with administration of the first chemotherapy dose of a chemotherapy block and continued until 24 hours after administration of the last chemotherapy dose of the block. Acute Phase - bands will be worn on each day of the chemotherapy course and for 24 hours after the last chemotherapy dose. Nausea severity during the acute phase of chemotherapy is defined as the maximum PeNAT (Pediatric Nausea Assessment Tool) score observed during each 24 hour period. The possible scores for the pediatric nausea assessment tool are no nausea, mild nausea, moderate nausea, severe nausea. Only patients who contributed at least 1 PeNAT score during the acute phase were included. The duration of the acute phase varied with chemotherapy regimen, according to study design.
Time Frame: Each day of Chemotherapy course. Maximum of 7 days
Population: The overall number of patients analyzed is 83 for Arm I and 82 for Arm II. Patients analyzed include the total number of patients that reported at least 1 PeNAT (Pediatric Nausea Assessment Tool) score on that day. The duration of the acute phase varied with chemotherapy regimen, according to study design. The number of patients receiving chemotherapy for longer than 3 days diminished each day, so days 4-7 were collapsed and considered a single day.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands
Number analyzed (Participants) | 83 | 82
Participants
  Day 1: number analyzed (Participants) | 82 | 80
  Day 1: No Nausea | 37 | 41
  Day 1: Mild Nausea | 17 | 8
  Day 1: Moderate Nausea | 16 | 19
  Day 1: Severe Nausea | 12 | 12
  Day 2: number analyzed (Participants) | 80 | 80
  Day 2: No Nausea | 17 | 15
  Day 2: Mild Nausea | 23 | 27
  Day 2: Moderate Nausea | 24 | 20
  Day 2: Severe Nausea | 16 | 18
  Day 3: number analyzed (Participants) | 70 | 64
  Day 3: No Nausea | 13 | 16
  Day 3: Mild Nausea | 19 | 17
  Day 3: Moderate Nausea | 18 | 21
  Day 3: Severe Nausea | 20 | 10
  Days 4-7: number analyzed (Participants) | 50 | 43
  Days 4-7: No Nausea | 13 | 16
  Days 4-7: Mild Nausea | 10 | 12
  Days 4-7: Moderate Nausea | 11 | 10
  Days 4-7: Severe Nausea | 16 | 5

2. Secondary Outcome: Efficacy of Treatment on CIN During Delayed Phase of Chemotherapy
Description: CIN = Chemotherapy-Induced Nausea. The delayed phase began at the end of the acute phase and continued until the first chemotherapy dose of the next chemotherapy block. Delayed Phase - Bands will continue to be worn for a maximum of 7 days or until the next chemotherapy cycle starts, whichever comes first. Nausea severity is defined as the maximum PeNAT (Pediatric Nausea Assessment Tool) score observed during each 24 hour period. The possible scores for the pediatric nausea assessment tool are no nausea, mild nausea, moderate nausea, severe nausea. Only patients who contributed at least 1 PeNAT score during the delayed phase were included.
Time Frame: Maximum of 7 days after Acute Phase
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands
Number analyzed (Participants) | 83 | 82
Participants
  Day 1: number analyzed (Participants) | 75 | 68
  Day 1: No Nausea | 27 | 27
  Day 1: Mild Nausea | 19 | 15
  Day 1: Moderate Nausea | 19 | 13
  Day 1: Severe Nausea | 10 | 13
  Day 2: number analyzed (Participants) | 67 | 62
  Day 2: No Nausea | 28 | 25
  Day 2: Mild Nausea | 15 | 20
  Day 2: Moderate Nausea | 15 | 12
  Day 2: Severe Nausea | 9 | 5
  Day 3: number analyzed (Participants) | 65 | 61
  Day 3: No Nausea | 28 | 33
  Day 3: Mild Nausea | 21 | 14
  Day 3: Moderate Nausea | 12 | 7
  Day 3: Severe Nausea | 4 | 7
  Days 4-7: number analyzed (Participants) | 56 | 51
  Days 4-7: No Nausea | 19 | 28
  Days 4-7: Mild Nausea | 13 | 13
  Days 4-7: Moderate Nausea | 14 | 3
  Days 4-7: Severe Nausea | 10 | 7

3. Secondary Outcome: Comparison of Control of CIV During the Acute and Delayed Phase of Chemotherapy
Description: CIV = Chemotherapy-Induced Vomiting. Total Duration of Study includes both acute and delayed phases. Acute Phase - bands will be worn on each day of the chemotherapy course and for 24 hours after the last chemotherapy dose. Delayed Phase - Bands will continue to be worn for a maximum of 7 days or until the next chemotherapy cycle starts, whichever comes first. A breakthrough antiemetic agent is defined as a medication that is administered or taken in order to relieve or treat (rather than prevent) nausea or vomiting. An antiemetic agent that is prescribed and/or administered on an "as needed" basis is considered to be a breakthrough antiemetic. Complete CIV Control during the acute and delayed phases is defined as no emetic episodes and no breakthrough anti-emetic agents administered during the phase of interest. Partial CIV Control is defined as 1 or 2 emetic episodes in any 24 ho
Time Frame: Maximum of 14 days
Population: The overall number of participants analyzed is 83 participants in Arm I and 82 participants in Arm II. In the acute phase, 165 patients provided at least 1 PeNAT (Pediatric Nausea Assessment Tool) score. In the delayed phase, 144 patients contributed at least 1 PeNAT score.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands
Number analyzed (Participants) | 83 | 82
Participants
  Acute Phase: Complete CIV Control | 17 | 19
  Acute Phase: Partial CIV Control | 43 | 48
  Acute Phase: Failed CIV Control | 23 | 15
  Delayed Phase: number analyzed (Participants) | 75 | 69
  Delayed Phase: Complete CIV Control | 35 | 31
  Delayed Phase: Partial CIV Control | 29 | 28
  Delayed Phase: Failed CIV Control | 11 | 10

ADVERSE EVENTS:
Time Frame: First application of wrist bands through 8 days after administration of the last chemotherapy dose of the cisplatin-containing course.
Description: Adverse events could spontaneously be communicated by the patient/family and/or elicited via the Final Questionnaire.
Arm/Group | Arm I- Real Acupressure Bands | Arm II- Placebo Acupressure Bands
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/83 | 0/82
Other Adverse Events (participants affected / at risk) | 0/83 | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No